CLINICAL TRIAL: NCT05869838
Title: Collecting Real-world Data on Endoscopic and Histopathological Outcomes of Screening and Surveillance Colonoscopies for the Development of a CAD (Computer Aided Detection) System: a Prospective, Multicenter, Post-market Investigation
Brief Title: A Clinical Study on Endoscopic and Histopathological Outcomes of Screening and Surveillance Colonoscopies
Acronym: CODACO
Status: Recruiting | Type: Observational
Sponsor: Olympus Europe SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-001
Record Dates: First submitted 2023-05-09; First posted 2023-05-22 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Colonic Polyp
MeSH Terms: conditions — Colonic Polyps | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Colonoscopy — Screening or surveillance colonoscopy

SUMMARY:
The objective of this study is to collect colonoscopy data for use in the development and testing of artificial intelligence (AI) devices for colonoscopies.

DETAILED DESCRIPTION:
The primary objective of this study is to collect colonoscopy data for use in the development and performance evaluation of AI devices. The data will be collected during routine colonoscopy procedures. Biopsy or resection will be performed if needed and all specimens will be sent for histopathological examination. The histopathological results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients who have signed a written consent form from their voluntary decision after receiving thorough explanation on this study and fully understanding the explanation prior to participation in the study
* Patients who plan to receive colonoscopy procedure and meet any of the following conditions: Colon cancer screening, post-polypectomy surveillance, patients who are advised by a physician to take a colonoscopy exam

Exclusion Criteria:

* Patients for whom endoscopic submucosal dissection is planned
* Patients for whom polypectomy is difficult to perform due to antithrombotic therapy received etc.
* Patients who have to receive an urgent colonoscopy procedure
* Patients who underwent total colectomy of the large intestine
* Patients who are judged by a physician to be contraindicated for colonoscopy procedures
* Patients who have participated in another clinical study within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing screening or surveillance colonoscopy
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Videos and still images of the colonoscopy | during the procedure
  Narrow band imaging (NBI) images and white-light images, video recordings of the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sofía Parejo Carbonell, Principal Investigator — Hospital Universitario Ramón y Cajal
Locations (3):
- End- und Dickdarmzentrum Hannover, Hanover, Germany
- Hospital Universitario Ramón y Cajal, Madrid, Spain
- Ersta Hospital Stockholm, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No